CLINICAL TRIAL: NCT03771911
Title: Quality of Cardiopulmonary Resuscitation Guided by AED vs Telephone-assistance
Acronym: QRCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bionorte (Other)
Collaborators: University of the Basque Country (UPV/EHU) (Other); Osakidetza (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: QRCP
Record Dates: First submitted 2018-12-02; First posted 2018-12-11 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-05

CONDITIONS: Cardiopulmonary Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AED guided (Other): Laypeople will be guided by an Automatic External Defibrillator's (AED) voice instructions during the cardiopulmonary resuscitation.
  No other help is available.
  Interventions: Device: AED
- Telephone guided (Other): Laypeople will be guided by telephone assistance (from an Emergency Call Center) during the cardiopulmonary resuscitation.
  AED voice instructions are also available.
  Interventions: Device: AED; Device: Telephone

INTERVENTIONS:
Device: AED — Instructions provided by an AED
Device: Telephone — Instructions provided by emergency Call Center (telephonically) with the help of an AED.
  Arms: Telephone guided

SUMMARY:
The aim of this research is to evaluate and to compare the quality of cardiopulmonary resuscitation (CPR) among untrained laypeople under two different scenarios: automated external defibrillator (AED) guided CPR or dispatcher-assisted CPR. Secondarily, to evaluate the quality of the dispatcher-assisted instructions provided from the emergency call center.

DETAILED DESCRIPTION:
A simulation study will beperformed. 42 volunteers selected by non-probabilistic sampling will be randomized in two scenarios of cardiac arrest on mannequin: (A) AED-guided CPR and (T) dispatcher-assisted CPR. Simulations last 9 minutes. The quality of CPR will be evaluated by metric monitoring of the chest compressions and timing of actions. A peer's content analysis of the telephone instructions will be performed using a checklist.

ELIGIBILITY:
Inclusion Criteria:

* untrained laypeople
* Volunteers

Exclusion Criteria:

* Pregnants, leg/arm injuried people, chronic back pain.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-05-27 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary resuscitations strated | 9 minutes
  nº of CPR strated by bystander

SECONDARY OUTCOMES:
Chest compressions rate | 9 minutes
  Chest compression/minute
Chest compressions depth/recoil | 9 minutes
  % os chest compressions with correct depth/recoil
Time under CPR | 8 minutes
  % of time applying chest compressions
Hands on chest | 9 minutes
  % of chest compressions with a correct position of hands

CONTACTS AND LOCATIONS:
Overall Officials: Irrintzi Fernández-Aedo, PhD, Study Chair — University of the Basque Country (UPV/EHU); Gorka Vallejo-De la Hoz, PhD, Study Chair — Osakidetza; Alejandro Etayo-Sancho, RN, Study Chair — Ambuiberica; Asier Alonso-Pinillos, RN, Study Chair — Osakidetza; Sendoa Ballesteros-Peña, PhD, Study Director — Osakidetza
Locations (1):
- Hospital de Basurto, Bilbao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: No